CLINICAL TRIAL: NCT06869187
Title: A Phase 2 Open-label Study of the Effect of Adjunctively Administered ABX-002 in Adults With Bipolar Disorder Experiencing an Episode of Depression
Brief Title: Study of ABX-002 for the Adjunctive Treatment of Depressive Episodes Associated With Bipolar Disorder in Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Autobahn Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX-002-2002
Record Dates: First submitted 2025-02-18; First posted 2025-03-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Bipolar Disorder Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABX-002 + at least one mood stabilizer and/or single second-generation antipsychotic (SGA) (Experimental): Participants will continue all medications intended to treat the current episode of depression for the duration of the study in addition to ABX-002
  Interventions: Drug: ABX-002
- No Treatment + Imaging Sessions (No Intervention): Healthy Volunteers will not receive any study treatment as their only assessment is 2 imaging sessions (baseline and retest)

INTERVENTIONS:
Drug: ABX-002 — ABX-002 oral solution in 1-mL cyclic olefin polymer prefilled syringes, taken on an empty stomach first thing in the morning followed by 240 mL (8 oz) of water.
  Arms: ABX-002 + at least one mood stabilizer and/or single second-generation antipsychotic (SGA)

SUMMARY:
The goal of this clinical trial is to learn if ABX-002 added to participants' existing treatment(s) can improve clinical symptoms of depression and to learn about potential effects on brain chemistry that may correlate with antidepressive effects.

This is a single treatment arm, open-label, Phase 2 study of ABX-002 in up to30 adults with bipolar depression. A subset of these participants will undergo brain imaging. Five healthy volunteer participants will also be enrolled and receive no drug treatment, undergoing 2 imaging sessions to confirm instrument and test - retest method reliability control.

For bipolar disorder participants who are experiencing an episode of depression, the study will include 4 study periods:

1. Screening Period of up to 5 weeks
2. 6-week Treatment Period
3. 2-week post dose Safety Follow-up Period.
4. 6-month postdose targeted safety follow-up period

For healthy volunteers, the study will include 2 study periods:

1. Screening Period of up to 3 weeks
2. Imaging Period of up to 3 weeks.

ELIGIBILITY:
Inclusion Criteria (For Bipolar Disorder Depression Patients):

* Current diagnosis of bipolar disorder for at least 2 years
* DSM-5-TR criteria for bipolar disorder based on Structured Clinical Interview for the DSM-5 - Clinical Trials Version (SCID-5-CT) at Screening
* Has a current depressive episode with or without mixed features, but not psychotic features, with duration ≥ 6 weeks and ≤ 24 months
* 17-item Hamilton Rating Scale for Depression total score ≥ 22 at Screening and Baseline
* Young Mania Rating Scale total score ≤ 12 at Screening and Baseline
* For participants who will undergo brain imaging: Able to undergo imaging sessions using Magnetic Resonance Spectroscopy/Imaging with no history of aborted scanning due to anxiety, claustrophobia, or unable to scan due to an incompatible implant/device
* Taking at least one mood stabilizer (e.g., lithium, valproate, lamotrigine) and/or second-generation antipsychotic (SGA, atypical antipsychotic). All medications intended to treat the current episode of depression should be at an adequate and stable dose for ≥ 6 weeks prior to screening.

Exclusion Criteria (For Bipolar Disorder Depression Patients):

* History of > 4 manic, hypomanic, or depressive episodes within a one-year period (rapid cycler; DSM-5-TR) in the last 2 years
* History of schizophrenia or schizoaffective disorder (DSM-5-TR) or a psychotic disorder unrelated to bipolar disorder
* Concurrent or history of active symptoms within the past 2 years of obsessive-compulsive disorder, or posttraumatic stress disorder, according to DSM-5-TR criteria
* Diagnosis of a personality disorder (DSM-5-TR)
* Evident risk of suicide at Screening or Baseline
* Inadequate response to more than 2 second-generation antipsychotic treatments (including their current treatment) in their current episode of depression in bipolar disorder despite an adequate dose and duration (> 6 weeks at approved or standard of care doses)
* Received any course of deep brain stimulation in participant's lifetime or plans to receive deep brain stimulation during the study
* Treatment with electroconvulsive therapy (for psychiatric/therapeutic purposes) or repetitive transcranial magnetic stimulation, or treatment with ketamine or esketamine for the current episode and received any of those treatments within 12 months prior to Screening
* Started new psychotherapy or had a change in the intensity of psychotherapy within 6 weeks before Screening
* Prior use of psychedelics for the treatment of depression
* Refusal to abstain from consumption of excessive amounts of alcohol during the study
* History of uncontrolled, clinically significant neurological (including prior cerebrovascular accident [stroke] or chronic seizures), cardiovascular, gastrointestinal, respiratory, renal, hepatic, immunological, hematological, endocrine (including uncontrolled diabetes), or other medical disorder, including cancer
* Current use of high dose (> 4 mg/day lorazepam equivalents) benzodiazepine anxiolytic and/or hypnotic medication
* Cannabinoids (marijuana, cannabis, tetrahydrocannabinol [THC], cannabidiol [CBD]) in any form or use frequency.
* History or presence of cataract on ophthalmic examination (including slit-lamp), glaucoma, inflammatory eye disease prior ophthalmic surgical procedures or laser surgery in either eye.

Inclusion Criteria (For Healthy Volunteers):

* In good health, based on medical history, physical examination (including neurological examination), vital sign measurements, and laboratory safety tests obtained at the Screening Visit
* Able to undergo imaging sessions using Magnetic Resonance Spectroscopy/Imaging, with no history of aborted scanning due to anxiety, claustrophobia, or an incompatible implant/device

Exclusion Criteria (Healthy Volunteers):

* Mentally or legally incapacitated, has significant emotional problems at the time of the Screening Visit, or is expected to have potential for mental incapacitation during the conduct of the study
* History of any illness (including psychiatric illness)
* Participation in an investigational drug or device study where last dosing of previous drug is within 30 days
* Prior use of psychedelics within the past year
* Refusal to abstain from consumption of excessive amounts of alcohol during the study
* Cannabinoids (marijuana, cannabis, tetrahydrocannabinol [THC], cannabidiol [CBD]) in any form or use frequency are not allowed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Change from baseline for 17-item Hamilton Rating Scale for Depression (HAMD-17) | Weeks 6
  HAMD-17 is a clinician-based assessment of depressive symptoms. Higher scores indicate worse symptoms. A score of 0-9 is generally accepted to be within the normal range (or in clinical remission), while a score of greater than 17 indicates moderate to severe depression symptoms.

SECONDARY OUTCOMES:
Correlation of change from baseline in the anterior cingulate cortex (ACC) nucleoside triphosphate/inorganic phosphate (NTP/Pi) concentrations with percentage change in Hamilton Depression Rating Scale (HAMD)-17 | Week 6
  Utilizing 31P-Magnetic Resonance Spectroscopy (31P-MRS), a magnetic resonance imaging (MRI) method that measures high-energy phosphates in the brain
Correlation of change from Baseline in the anterior cingulate cortex (ACC) phosphocreatine/inorganic (PCr/Pi) concentration with percentage change in Hamilton Depression Rating Scale (HAMD)-17 | Week 6
  Utilizing 31P-Magnetic Resonance Spectroscopy (31P-MRS), a magnetic resonance imaging (MRI) method that measures high-energy phosphates in the brain
Change from baseline for 29-item Hamilton Rating Scale for Depression (HAMD-29) | Weeks 6
  HAMD-29 is a clinician-based assessment of depressive symptoms. Higher scores indicate worse symptoms. A score of 0-7 is generally accepted as not depressed, 8-16 indicates mild depression, 17-23 indicates moderate depression, and 24 and above indicates severe depression.
Change from baseline in 6-item Hamilton Rating Scale for Depression (HAMD-6) | Weeks 6
  Six-item scale used to assess the core symptoms of depression. HAMD-6 is a shorter version of HAMD-17. The higher the total score the more severe the depression.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Autobahn Site #213, Walnut Creek, California
  - Autobahn Site #201, Cromwell, Connecticut
  - Autobahn Site #210, Hartford, Connecticut
  - Autobahn Site #212, Miami, Florida
  - Autobahn Site #215, Chicago, Illinois
  - Autobahn Site #216, Worcester, Massachusetts
  - Autobahn Site #208, Cherry Hill, New Jersey
  - Autobahn Site #209, Hamilton, New Jersey
  - Autobahn Site #205, Marlton, New Jersey
  - Autobahn Site #203, Brooklyn, New York
  - Autobahn Site #207, New York, New York
  - Autobahn Site #211, New York, New York
  - Autobahn Site #202, New York, New York
  - Autobahn Site #204, Staten Island, New York
  - Autobahn Site #214, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No